CLINICAL TRIAL: NCT06546202
Title: Real-World Pharmacological Treatment Pattern of Neuropathic Pain in China: A Retrospective, Database, Multi-center Study (ReTARdant)
Brief Title: Real-World Pharmacological Treatment Pattern of Neuropathic Pain in China
Status: Completed | Type: Observational
Sponsor: Daiichi Sankyo (Industry)
Collaborators: Daiichi Sankyo Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: DS5565-0001-NIS-MA
Record Dates: First submitted 2024-08-06; First posted 2024-08-09 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Diabetic Peripheral Neuropathic Pain; Chemotherapy-induced Peripheral Neuropathy; Neuropathic Pain
Keywords: Diabetic peripheral neuropathic pain; Chemotherapy-induced peripheral neuropathy; Neuropathic pain; Treatment pattern
MeSH Terms: conditions — Neuralgia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Diabetic peripheral neuropathic pain: Participants who have been diagnosed with diabetic peripheral neuropathic pain and presented with pain symptoms.
  Interventions: Other: No Drug
- Chemotherapy-induced peripheral neuropathy: Participants who have chemotherapy-induced peripheral neuropathy regardless of the presence of pain symptoms.
  Interventions: Other: No Drug

INTERVENTIONS:
Other: No Drug — This is an non-interventional, observational study. No drug was administered during this study.

SUMMARY:
The aim of this study is to investigate the pharmacological treatment pattern among patients with diabetic peripheral neuropathic pain (DPNP) and chemotherapy-induced peripheral neuropathy (CIPN) in China.

DETAILED DESCRIPTION:
Diabetic peripheral neuropathic pain (DPNP) and chemotherapy-induced peripheral neuropathy (CIPN) are common subtypes of neuropathic pain. The treatment pattern, subsequent medication usage, and adherence information of medication among these patients are still not clear. There is also an unmet need for the use of relevant analgesic medications in this area. This real-world data study aims to understand patients' characteristics, clinical diagnosis and treatment patterns, medication adherence, real-world effectiveness among DPNP and CIPN patients in China and will explore the current unmet needs of DPNP and CIPN, in order to inform physicians' decision-making in clinical practice

ELIGIBILITY:
Participants who meet all the following criteria will be included in the DPNP cohort.

1. Participants were diagnosed with diabetic neuropathy and presented with the pain symptom between 1st January 2018 and 31st December 2021;
2. Participants received at least one targeted medication between 1st January 2018 and 31st December 2021;
3. Participants were ≥18 years on the index date;
4. Participants had at least one medical visit record within 12 months after the index date

Participants who meet any one of the following criteria will be excluded from the DPNP cohort.

(1) Participants were diagnosed with epilepsy, schizophrenia, or bipolar disorder before or on the index date

Participants who meet all the following criteria will be included in the CIPN cohort.

1. Participants had neuropathy that was induced by the chemotherapy between 1st January 2018 and 31st December 2021, regardless of the presence of pain symptoms;
2. Participants received at least one targeted medication between 1st January 2018 and 31st December 2021;
3. Participants were ≥18 years on the index date;
4. Participants had at least one medical visit record within12 months after the index date

Participants who meet any one of the following criteria will be excluded from the CIPN cohort.

1. Participants were diagnosed with epilepsy, schizophrenia, or bipolar disorder before or on the index date;
2. Participants had neuralgia or neuropathy caused by tumor metastasis or non-chemotherapy-induced factors (e.g., radiotherapy, myasthenia gravis syndrome, paraneoplastic syndrome, direct tumor invasion, local tissue compression, postoperative traumatic pain, immune therapy-related pain, comorbidity-induced pain, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study target population is eligible participants from general hospitals and oncology-specialized hospitals in several provinces and regions of China who were diagnosed with DPNP or CIPN between 1st January 2018 and 31st December 2021 and received the targeted medications.
Sampling Method: Non-Probability Sample
Enrollment: 1271 (Actual)
Dates: Start 2024-08-16 (Actual); Primary Completion 2025-07-18 (Actual); Study Completion 2025-07-18 (Actual)

PRIMARY OUTCOMES:
Proportion of participants receiving different treatment regimens (targeted medications or combinations) and related medication categories in participants with DPNP or CIPN | From index date up to 31st December 2022
  The treatment regimen will be evaluated and confirmed as monotherapy or combination therapy based on prescription records at each visit. Monotherapy is defined as participants only received one targeted medication. Combination therapy is defined as participants received more than one targeted medication at the same time.
Proportion of participants who discontinue/switch/add-on treatment and related medication categories in participants with DPNP or CIPN | From index date up to 31st December 2022
  Treatment discontinuation is defined as the time interval between two adjacent treatment regimens, or the time interval between the end of the last treatment regimen and the study end date (31st December 2022), or the time interval between the end of the last treatment regimen and the date of death is ≥90 days. Treatment switch is defined as the change of treatment regimen, either in monotherapy or in combination (exclude treatment add-on). Treatment add-on is defined as the addition of one or more targeted medications to an existing treatment regimen (monotherapy or combination therapy).
Proportion of participants who restarted treatment after discontinuation in participants with DPNP or CIPN | From index date up to 31st December 2022
  Among those who had discontinued treatment, the proportion of patients who received at least one targeted medication at the next visit will be assessed, where the treatment regimen containing the targeted medication includes the same treatment medication prior to discontinuation or a different treatment medication after treatment switch/add-on.
Duration of the current treatment in participants with DPNP or CIPN | From index date up to 31st December 2022
  Duration of the current treatment is defined as the time interval from the start date of a treatment to its end date. The end date of the treatment refers to its discontinuation date; for participants who did not experience a treatment discontinuation, the end date of treatment prescription is used.
Time to treatment add-on in participants with DPNP or CIPN | From index date up to 31st December 2022
  Time to treatment add-on is defined as the time interval between the end date of the current treatment regimen (including days covered by take-away medications) and the start date of the add-on treatment.

SECONDARY OUTCOMES:
Initial daily dose in participants with DPNP or CIPN | From index date up to 31st December 2022
  Initial daily dose is defined as the first prescribed daily dose of the targeted medications.
Maximum daily dose in participants with DPNP or CIPN | From index date up to 31st December 2022
  Maximum daily dose is defined as the maximum of the daily dose.
Time to the maximum daily dose in participants with DPNP or CIPN | From index date up to 31st December 2022
  Time to the maximum daily dose is defined as the time interval between the daily dose to the maximum daily dose.
Proportion of participants who underwent the daily dose change in participants with DPNP or CIPN | From index date up to 31st December 2022
  Proportion of participants who underwent the daily dose change is defined as the proportion of participants who underwent the dose changes from the initial daily dose to 2 weeks, 4 weeks and 6 weeks, respectively.

CONTACTS AND LOCATIONS:
Locations (10):
- China (10):
  - China-Japan Friendship Hospital, Beijing
  - Beijing Hospital, Beijing
  - Beijing Cancer Hospital, Beijing
  - The First Affiliated Hospital of Dalian Medical University, Dalian
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou
  - Sun Yat-Sen University Cancer Center, Guangzhou
  - Zhejiang Provincial People's Hospital, Hangzhou
  - Cancer Hospital of Shandong First Medical University (Shandong Cancer Institute, Shandong Cancer Hospital), Jinan
  - Liaoning Cancer Hospital & Institute, Shenyang
  - Tongji Hospital Tongji Medical College of Hust, Wuhan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pan Q, Zhai X, Wang H, Du J, Shi Y, Yu X, Yan S, Wu X, Li HH, Sun T, Guo L, Zhao J, Fan B. Real-World Pharmacological Treatment Pattern of Neuropathic Pain in China: A Retrospective, Database, Multicenter Study (ReTARdant) Protocol. Pain Ther. 2025 Oct;14(5):1611-1627. doi: 10.1007/s40122-025-00767-x. Epub 2025 Aug 11. PMID 40788612